CLINICAL TRIAL: NCT03441113
Title: Extended Access of Momelotinib for Subjects With Primary Myelofibrosis (PMF) or Post-polycythemia Vera or Post-essential Thrombocythemia Myelofibrosis (Post-PV/ET MF)
Brief Title: Extended Access of Momelotinib in Adults With Myelofibrosis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 219627; 2017-004350-42 (EudraCT Number); SRA-MMB-4365 (Other: Sierra Oncology, Inc.); 219627 (Other: GlaxoSmithKline)
Record Dates: First submitted 2018-02-15; First posted 2018-02-22 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Neoplasms; Post-polycythemia Vera Myelofibrosis (Post-PV MF); Primary Myelofibrosis (PMF); Post-essential Thrombocythemia Myelofibrosis (Post-ET MF)
MeSH Terms: conditions — Neoplasms; Primary Myelofibrosis | interventions — N-(cyanomethyl)-4-(2-((4-(4-morpholinyl)phenyl)amino)-4-pyrimidinyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: Study GS-US-352-0101 (Other): Participants will continue to receive the same dosage regimen as in the previous MMB study GS-US-352-0101 until MMB receives regulatory approval and is commercially available, or development of the product ceases.
  Interventions: Drug: MMB
- Cohort 2: Study GS-US-352-1214 (Other): Participants will continue to receive the same dosage regimen as in the previous MMB study GS-US-352-1214 until MMB receives regulatory approval and is commercially available, or development of the product ceases.
  Interventions: Drug: MMB
- Cohort 3: Study GS-US-352-1154 (Other): Participants will continue to receive the same dosage regimen as in the previous MMB study GS-US-352-1154 until MMB receives regulatory approval and is commercially available, or development of the product ceases..
  Interventions: Drug: MMB
- Cohort 4: Study SRA-MMB-301 (Other): Participants will continue to receive the same dosage regimen as in the previous MMB study SRA-MMB-301 until MMB receives regulatory approval and is commercially available, or development of the product ceases.
  Interventions: Drug: MMB

INTERVENTIONS:
Drug: MMB — Tablet(s) administered orally once daily
  Other Names: GS-0387; CYT387

SUMMARY:
The primary objective of this study is to provide extended access and assess long-term safety of momelotinib (MMB) in participants with primary myelofibrosis (PMF) or post-polycythemia vera or post-essential thrombocythemia myelofibrosis (Post-PV/ET MF) enrolled in studies GS-US-352-0101 (NCT01969838), GS-US-352-1214 (NCT02101268), GS-US-352-1154 (NCT02124746), SRA-MMB-301 who are currently receiving treatment with MMB (available as 50mg,100 mg, 150 mg and 200 mg tablets) and have not experienced progression of disease. The secondary objective is to assess overall survival (OS) and leukemia free survival (LFS) in all subjects.

ELIGIBILITY:
Key Inclusion Criteria:

* Currently enrolled in Studies GS-US-352-0101, GS-US-352-1214, GS-US-352-1154, or SRA-MMB-301
* Able to comprehend and willing to sign the informed consent form

Key Exclusion Criteria:

* Known hypersensitivity to MMB, its metabolites, or formulation excipients

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Had Access to, and Received the Intervention | Participants will be assessed every 12 weeks until discontinuation. Participation in this extended access study has been an average of approximately 8 months.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (212):
- United States (29):
  - IC Irvine Health, Orange, California
  - GSK Investigational Site, Stanford, California
  - Stanford Hospital and Clinics, Stanford, California
  - GSK Investigational Site, Aurora, Colorado
  - University of Colorado Cancer Center, Aurora, Colorado
  - GSK Investigational Site, Jacksonville, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - GSK Investigational Site, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Northwest Oncology & Hematology - Rolling Meadows, Rolling Meadows, Illinois
  - GSK Investigational Site, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - Dana-Farber Cancer Institute (DFCI), Boston, Massachusetts
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Rochester, Minnesota
  - Mayo Clinic - Department of Hematology, Rochester, Minnesota
  - Washington University School of Medicine Siteman Cancer Center, St Louis, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Hackensack, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - GSK Investigational Site, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Milwaukee, Wisconsin
  - Mayo Clinic Building - Phoenix, Milwaukee, Wisconsin
- Australia (12):
  - Icon Cancer Care Wesley, Hyde Park, Queensland
  - GSK Investigational Site, South Brisbane, Queensland
  - Flinders Medical Centre, Adelaide, South Australia
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Frankston, Victoria
  - Frankston Hospital, Frankston, Victoria
  - GSK Investigational Site, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - GSK Investigational Site, Parkville, Victoria
  - Peter MacCallum Cancer Centre, Parkville, Victoria
  - GSK Investigational Site, Perth, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Austria (4):
  - Ordensklinikum Linz Elisabethinen, Linz, Upper Austria
  - Medizinische Universität Wien, Vienna, Vienna
  - GSK Investigational Site, Linz
  - GSK Investigational Site, Vienna
- Belgium (8):
  - Algemeen Ziekenhuis Sint-Jan Brugge-Oostende - Campus Sint-Jan, Bruges, West-Vlaanderen
  - GSK Investigational Site, Antwerp
  - Ziekenhuis Netwerk Antwerpen Stuivenberg, Antwerp
  - GSK Investigational Site, Bruges
  - GSK Investigational Site, Leuven
  - Universitaire Ziekenhuis Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège Site Sart Tilman, Liège
  - GSK Investigational Site, Liège
- Bulgaria (7):
  - GSK Investigational Site, Pleven
  - UMHAT Dr. Georgi Stranski EAD, Pleven
  - GSK Investigational Site, Rousse
  - Multiprofile Hospital for Active Treatment Ruse, Rousse
  - GSK Investigational Site, Sofia
  - National Specialized Hospital for Active Treatment of Haematologic Diseases, Sofia
  - University Multiprofile Hospital for Active Treatment St. Ivan Rilski, Sofia
- Canada (5):
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - Research Institute of the McGill University Health Centre, Montreal, Quebec
  - Sir Mortimer B. Davis Jewish General Hospital, Montreal
  - Princess Margaret Cancer Centre, Toronto
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - GSK Investigational Site, Aalborg
  - GSK Investigational Site, Copenhagen
  - Gentofte Hospital, Herlev
- France (13):
  - Centre Hospitalier Le Mans, Le Mans, Pays de la Loire Region
  - GSK Investigational Site, Le Mans
  - CHRU Huriez Lille, Lille
  - GSK Investigational Site, Marseille
  - Institut Paoli Calmettes, Marseille
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pessac
  - Hôpital Haut-Lévêque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - GSK Investigational Site, Pierre-Bénite
  - GSK Investigational Site, Toulouse
  - Institut Universitaire du Cancer, Toulouse
  - Hopital Saint-Louis, Paris, Île-de-France Region
- Germany (14):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Aachen, North Rhine-Westphalia
  - Universitätsklinikum Aachen, Aachen, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Halle, Saxony-Anhalt
  - Universitätsklinikum Halle, Halle, Saxony-Anhalt
  - Universitätsklinikum Schleswig-Holstein - Campus Lübeck, Lübeck, Schleswig-Holstein
  - University Hospital of Cologne, Cologne
  - Universitätsklinikum Dresden, Dresden
  - Universitätsklinikum Leipzig, Leipzig
  - Johannes Gutenberg-Universität Mainz, Mainz
- Hungary (13):
  - Petz Aladár Egyetemi Oktató Kórház - Győr, Győr, Győr-Moson-Sopron
  - Szent Borbála Kórház, Tatabánya, Komárom-Esztergom
  - Dél-pesti Centrumkórház - Országos Hematológiai és Infektológiai Intézet, Budapest, Pest County
  - Szabolcs-Szatmár-Bereg Megyei Kórházak És Egyetemi Oktatókórház, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - GSK Investigational Site, Budapest
  - Semmelweis Egyetem I. sz. Belgyogyaszati Klinika, Hematologia, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Belgyogyaszati Klinika, Haematologiai Tanszek, Debrecen
  - GSK Investigational Site, Debrecen
  - GSK Investigational Site, Győr
  - GSK Investigational Site, Kaposvár
  - Somogy Megyei Kaposi Mor Oktató Kórház, Kaposvár
  - GSK Investigational Site, Nyíregyháza
  - GSK Investigational Site, Tatabánya
- Israel (10):
  - GSK Investigational Site, Afula
  - Emek Medical Center, Afula
  - Barzilai Medical Center, Hematology Institute, Ashkelon
  - GSK Investigational Site, Ashkelton
  - Carmel Medical Center, Haifa
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Jerusalem
  - Hadassh Medical Organization, Jerusalem
  - Meir Medical Center, Kfar Saba
  - GSK Investigational Site, Kfar Saba
- Italy (24):
  - GSK Investigational Site, Rionero in Vulture (Pz), Basilicate
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Bologna, Emilia-Romagna
  - Azienda Ospedaliero - Universitaria Careggi, Florence, Florence
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Monza (MB), Lombardy
  - Azienda Socio Sanitaria Territoriale Monza - Ospedale San Gerardo, Monza, Monza E Brianza
  - Azienda Ospedaliera Ospedali Riuniti Marche Nord, Pesaro, Pesaro E Urbino
  - GSK Investigational Site, Turin, Piedmont
  - GSK Investigational Site, Torino, Trentino-Alto Adige
  - Azienda Ospedaliero-Universitaria Citta della Salute e della Scienza di Torino, Torino, Turin
  - Azienda Ospedaliera Ordine Mauriziano di Torino, Torino, Turin
  - GSK Investigational Site, Florence, Tuscany
  - GSK Investigational Site, Verona, Veneto
  - Azienda Ospedaliero Universitaria di Bologna Policlinico Sant'Orsola-Malpighi, Bologna
  - Azienda Ospedaliera Universitaria San Martino, Genova
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - GSK Investigational Site, Pesaro
  - IRCCS Centro di Riferimento Oncologico di Basilicata, Potenza
  - GSK Investigational Site, Roma
  - Umberto I - Policlinico di Roma, Roma
  - Ospedale Policlinico Giambattista Rossi Borgo Roma, Verona
- Netherlands (2):
  - Maastricht University Medical Centre, Maastricht, Limburg
  - GSK Investigational Site, Maastricht
- Poland (14):
  - Szpital Wojewódzki w Opolu, Opole, Opole Voivodeship
  - Szpital Specjalistyczny w Brzozowie Podkarpacki Osrodek Onkologiczny im. Ks. B. Markiewicza, Brzozów, Podkarpacki
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Pomoskie
  - GSK Investigational Site, Brzozów
  - GSK Investigational Site, Chorzów
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Zespól Szpitali Miejskich, Chorzów
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lublin
  - Samodzielny Publiczny Szpital Kliniczny nr 1 w Lub, Lublin
  - Szpital Uniwersytecki w Krakowie, Oddzial Kliniczny Hematologii, Małogoskie
  - GSK Investigational Site, Opole
  - GSK Investigational Site, Poznan
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej MSWiA w Poznaniu im. Ledwika Bierkowskiego, Poznan
- Romania (11):
  - GSK Investigational Site, Brasov
  - Policlinica de Diagnostic Rapid SA, Brasov
  - GSK Investigational Site, Bucharest
  - Spitalul Clinic Coltea, Bucharest
  - Institutul Clinic Fundeni, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - Institutul Oncologic Prof. Dr. Ion Chiricuţă, Cluj-Napoca
  - GSK Investigational Site, Craiova
  - Spitalul Clinic Municipal Filantropia Craiova, Craiova
  - GSK Investigational Site, Iași
  - Institutul Regional De Oncologie IASI, Iași
- Singapore (3):
  - GSK Investigational Site, Singapore
  - Singapore General Hospital, Singapore
  - Raffles Hospital, Singapore
- South Korea (9):
  - Inje University Haeundae Paik Hospital, Busan, Busan Gwang'yeogsi [Pusan-Kwangyokshi]
  - Kyungpook National University Hospital, Daegu, Daegu Gwang'yeogsi
  - Severance Hospital, Seoul, Seoul Teugbyeolsi [Seoul-T'ukpyolshi]
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Seoul
  - Samsung Medical Center, Seoul
  - Catholic University of Korea Seoul Saint Mary's Hospital, Seoul
  - Seoul National University Hospital, Seoul
- Spain (13):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - GSK Investigational Site, Barcelona
  - Institut Hospital del Mar d'Investigacions Mèdiques, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - GSK Investigational Site, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid
  - GSK Investigational Site, Majadahonda (Madrid)
  - Clínica Universidad de Navarra, Pamplona
  - GSK Investigational Site, Pamplona
  - GSK Investigational Site, Zaragoza
  - Hospital de Día Quirónsalud Zaragoza, Zaragoza
- Taiwan (7):
  - GSK Investigational Site, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - GSK Investigational Site, Taipei
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou Branch, Taoyuan District
  - GSK Investigational Site, Taoyuan District
- United Kingdom (10):
  - University Hospitals Bristol and Weston NHS Foundation Trust, Bristol, England
  - GSK Investigational Site, Airdrie, Lanarkshire
  - NHS Lanarkshire, Airdrie, Scotland
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, Cardiff
  - University Hospital of Wales, Cardiff
  - GSK Investigational Site, London
  - Imperial College Healthcare NHS Trust, London
  - GSK Investigational Site, Oxford
  - Oxford University Hospitals NHS Trust, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gerds AT, Verstovsek S, Vannucchi AM, Al-Ali HK, Lavie D, Kuykendall AT, Grosicki S, Iurlo A, Goh YT, Lazaroiu MC, Egyed M, Fox ML, McLornan D, Perkins A, Yoon SS, Gupta V, Kiladjian JJ, Granacher N, Lee SE, Ocroteala L, Passamonti F, Harrison CN, Oh S, Klencke BJ, Yu J, Donahue R, Kawashima J, Mesa R. Momelotinib versus danazol in symptomatic patients with anaemia and myelofibrosis previously treated with a JAK inhibitor (MOMENTUM): an updated analysis of an international, double-blind, randomised phase 3 study. Lancet Haematol. 2023 Sep;10(9):e735-e746. doi: 10.1016/S2352-3026(23)00174-6. Epub 2023 Jul 27. PMID 37517413
- [Derived] Verstovsek S, Mesa R, Gupta V, Lavie D, Dubruille V, Cambier N, Platzbecker U, Hus M, Xicoy B, Oh ST, Kiladjian JJ, Vannucchi AM, Gerds A, Egyed M, Mayer J, Sacha T, Kawashima J, Morris M, Huang M, Harrison C. Momelotinib long-term safety and survival in myelofibrosis: integrated analysis of phase 3 randomized controlled trials. Blood Adv. 2023 Jul 25;7(14):3582-3591. doi: 10.1182/bloodadvances.2022009311. PMID 37042865